CLINICAL TRIAL: NCT02200003
Title: Attention Bias Modification for Anxiety: A Randomized Control Trial With Biomarkers
Acronym: ABMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Tracy Dennis, Professor, Hunter College of The City University of New York
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1 SC MH 109349-01
Record Dates: First submitted 2014-07-21; First posted 2014-07-25 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Anxiety
Keywords: attention bias modification, anxiety, event-related potentials
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: RCT of Attention Bias Modification
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attention Bias Modification (Experimental): 640 Trials (20 minutes) four times over four weeks
  Interventions: Behavioral: attention bias modification for anxiety
- Sham Attention bias modification (Sham Comparator): 640 Trials (20 minutes) four times over four weeks
  Interventions: Behavioral: attention bias modification for anxiety

INTERVENTIONS:
Behavioral: attention bias modification for anxiety

SUMMARY:
Computer-based attention bias modification treatment (ABMT), which is brief, cost-effective, and easy to administer, targets a key mechanism in pathological anxiety - the threat bias, or exaggerated attention feared or threatening stimuli. It remains unclear how and for whom ABMT is effective, limiting clinical translation. The proposed research involves an RCT using a highly sensitive measure of neurocognitive functioning, scalp-recorded event-related potentials (ERPs), to delineate key mechanisms of an emerging treatment for anxiety. Researchers will recruit 90 anxious participants to engage in the study and pursue the following three specific aims: Aim 1 will examine relations between neural and behavioral responses to threat prior to ABMT. Aim 2 will examine the effects of ABMT on ERPs to threat, threat bias, and anxiety. Aim 3 will examine relations between ERP responses to threat and reductions in threat bias and anxiety. Researchers will test whether post-training neural changes, specified in Aim 2, are associated with reductions in behavioral threat bias and anxiety severity. Researchers will also explore whether ERP measures of greater attention capture and/or reduced control of attention to threat at baseline predict treatment response, helping identify which patients will benefit most from ABMT. Through the innovative combination of a highly sensitive neurocognitive measure and an RCT design, this study aims to delineate core neurocognitive responses to threat as mechanisms in the remediation of anxiety. Confirmation of study hypotheses would, ultimately, accelerate the pace of development of more biologically-informed, accessible, and targeted interventions for anxiety.

DETAILED DESCRIPTION:
Anxiety disorders are the most common psychiatric diagnosis, affecting as many as 29% of people during their lifetime. In addition to the devastating personal cost of anxiety, the yearly economic cost to society has been estimated to be around $46.6 billion in the U.S. Empirically-based treatments for anxiety have improved in recent years, but barriers to access, side effects, and high remission rates (~50%) suggest the need for complementary treatments. Computer-based attention bias modification treatment (ABMT), which is brief, cost-effective, and easy to administer, targets a key mechanism in pathological anxiety - the threat bias, or exaggerated attention feared or threatening stimuli. Two decades of research show that reducing threat bias via computerized ABMT also reduces anxiety severity at levels comparable to gold-standard treatments. Despite its promise, no randomized clinical trials (RCTs) have evaluated specific mechanisms underlying ABMT's effects on anxiety, nor identified predictors of treatment response. Therefore, it remains unclear how and for whom ABMT is effective, limiting clinical translation. This study is a randomized clinical trial using a highly sensitive measure of neurocognitive functioning to delineate key mechanisms of an emerging treatment for anxiety. Specifically, the study will use scalp-recorded event-related potentials (ERPs) to elucidate neurocognitive processes implicated in attention bias modification treatment (ABMT) and to predict treatment response. Researchers will recruit 90 anxious patients to engage in the study and pursue the following three specific aims: Aim 1 will examine relations between neural and behavioral responses to threat prior to ABMT. Researchers will test whether greater behavioral threat bias is associated with ERP responses indicating greater attention capture by threat (larger P1 and P2 ERPs), and reduced top-down control of attention to threat (smaller N2, N2pc, P3 ERPs). Aim 2 will examine the effects of ABMT on ERPs to threat, threat bias, and anxiety. Analyses will focus on whether ABMT relative to placebo training will result in greater reductions in automatic attention capture and/or controlled attention to threat measured via ERPs. Aim 3 will examine relations between ERP responses to threat and reductions in threat bias and anxiety. Researchers will test whether post-training neural changes, specified in Aim 2, will be associated with reductions in behavioral threat bias and anxiety severity. These predicted relations,together with those tested in Aim 2a, support the utility of these ERPs as neural markers for the specific cognitive processes underlying ABMT efficacy. Researchers will also explore whether ERP measures of greater attention capture and/or reduced control of attention to threat at baseline predict treatment response, helping identify which patients will benefit most from ABMT. Through the innovative combination of a highly sensitive neurocognitive measure and an RCT design, this proposal aims to delineate core neurocognitive responses to threat as mechanisms in the remediation of anxiety. Confirmation of study hypotheses would, ultimately, accelerate the pace of development of more biologically-informed, accessible, and targeted interventions for anxiety.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit ninety adults with moderate to severe symptoms of anxiety between the ages of 21 and 40, with an equal balance of males and females.

Exclusion Criteria:

* Exclusion criteria include current or past episodes of disorders that include psychotic features (e.g., mania, schizophrenia, etc.,), suicidal intent, substance dependence, changes in pharmacological treatments during the 12 weeks prior to study entry, any concurrent psychotherapy, and serious medical illness.
* Other current and/or past Axis I diagnoses will not be excluded, but will be tracked.
* Given high rates of co-morbidity with anxiety, depressive symptoms will also be measured to assess impact on findings.
* To ensure understanding of the protocol, other exclusion criteria include inability to read, inability to complete assessments (i.e., severely impaired), and lack of English language comprehension.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in anxiety severity - immediate post intervention | Change in anxiety severity will be assessed five weeks after the baseline assessment
  Diagnostic interview using anxiety disorder modules only (MINI) and anxiety/impairment severity rating
Change in threat bias | Change in threat bias will be assessed five weeks after the baseline assessment
  RT-based measures of facilitated attention to threat (e.g., dot probe)
Change in anxiety severity - four-month follow-up | Change in anxiety severity will be assessed four months after the post-intervention assessment - a total of five months, one week from the baseline assessment
  Diagnostic interview using anxiety disorder modules only (MINI) and anxiety/impairment severity rating

SECONDARY OUTCOMES:
Change in neural responses to threat | Change in neural responses to threat will be assessed five weeks after the baseline assessment
  Scalp-recorded event-related potential measures (P1, P2, N2, P3) in response to threat stimuli
Change in behavioral stress reactivity | Change in behavioral stress reactivity will be assessed five weeks after the baseline assessment
  Observed and subjective feelings of stress and anxiety during the Trier Social Stress Test
Change in physiological measures of stress reactivity | Change in physiological stress reactivity will be assessed five weeks after the baseline assessment
  Heart rate and skin conductance during the Trier Social Stress Test

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Dennis, Ph.D., Principal Investigator — Hunter College of The City University of New York
Locations (1):
- Hunter College of the City University of New York, New York, New York, United States